CLINICAL TRIAL: NCT05011305
Title: A Phase 2b, Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Saroglitazar Magnesium in Subjects With Nonalcoholic Steatohepatitis and Fibrosis
Brief Title: Saroglitazar Magnesium for the Treatment of Nonalcoholic Steatohepatitis With Fibrosis
Acronym: NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SARO.20.002
Record Dates: First submitted 2021-07-11; First posted 2021-08-18 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Steatohepatitis; Fibrosis
Keywords: Saroglitazar Magnesium; Nonalcoholic Steatohepatitis; NASH; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — saroglitazar

STUDY DESIGN:
Intervention Model Description: 180 subjects randomized in a 1:1:1 ratio to Saroglitazar 2 mg, Saroglitazar 4 mg or Placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saroglitazar Magnesium 2 mg (Experimental): Saroglitazar Magnesium 2 mg tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment.
  Interventions: Drug: Saroglitazar Magnesium 2 mg
- Saroglitazar Magnesium 4 mg (Experimental): Saroglitazar Magnesium 4 mg tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment.
  Interventions: Drug: Saroglitazar Magnesium 4 mg
- Placebo (Placebo Comparator): Placebo tablet orally administered once daily in the morning before breakfast without food, for the duration of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saroglitazar Magnesium 2 mg — Patients randomly assigned to this group will receive Saroglitazar Magnesium 2 mg tablet orally once daily in the morning before breakfast without food, for the duration of treatment.
  Other Names: Investigational Product
  Arms: Saroglitazar Magnesium 2 mg
Drug: Saroglitazar Magnesium 4 mg — Patients randomly assigned to this group will receive Saroglitazar Magnesium 4 mg tablet orally once daily in the morning before breakfast without food, for the duration of treatment.
  Other Names: Investigational Product
  Arms: Saroglitazar Magnesium 4 mg
Drug: Placebo — Patients randomly assigned to this group will receive Placebo tablet orally once daily in the morning before breakfast without food, for the duration of treatment.
  Other Names: Comparator Agent
  Arms: Placebo

SUMMARY:
Saroglitazar Magnesium for the Treatment of Nonalcoholic Steatohepatitis

DETAILED DESCRIPTION:
A Phase 2b, Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Saroglitazar Magnesium in Subjects with Nonalcoholic Steatohepatitis and Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 75 years of age, both inclusive at screening.
* BMI ≤45 kg/m²
* Histological confirmation of NASH with liver fibrosis by central pathologist on a diagnostic liver biopsy with a NAS ≥4 with at least one-point score in each of the three components of the NAFLD activity score [NAS] (steatosis scored 0-3, ballooning degeneration scored 0-2, and lobular inflammation scored 0-3) and NASH by pattern recognition Note: The biopsy must not have been performed more than 24 weeks before randomization.
* The subjects must have a stable body weight (no more than 5% change) between the time of biopsy and randomization.
* Fibrosis stage 2 and 3, according to the NASH CRN fibrosis staging, reported by central pathologist.
* If the subjects have type 2 diabetes mellitus, then it must be moderately controlled with HbA1c ≤ 9.5% and on a stable dose of permitted anti-diabetic medication for at least 90 days before screening until randomization.
* If the subjects are taking vitamin E > 400 IU/day, then it must be on a stable dose for at least 24 weeks prior to screening or, if a historical biopsy is used, at least 24 weeks prior to baseline liver biopsy until randomization.
* Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

* Consumption of >2 units of alcohol per day (>14 units per week) if male and >1 units of alcohol per day (>7 units per week) if female for at least 12 consecutive weeks within 5 years before screening (Note: 1 unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor)
* History or presence of other concomitant liver diseases at screening:

  1. Chronic hepatitis B (HBV) or hepatitis C virus (HCV) infection (However, If the subject has been treated for the HCV infection and has been cured at least 5 years from screening, such subjects can be enrolled in the study)
  2. Primary biliary cholangitis (PBC)
  3. Primary sclerosing cholangitis (PSC)
  4. Definite autoimmune liver disease or overlap syndrome
  5. Alcoholic liver disease
  6. Hemochromatosis
  7. Wilsons disease
  8. Alpha-1 antitrypsin deficiency
* Subject with known cirrhosis, either based on histology, clinical criteria or any non-invasive diagnostic modality, within 24 weeks prior to the randomization.
* Evidence of portal hypertension (low platelet count, esophageal varices, ascites, history of hepatic encephalopathy, splenomegaly) at screening.
* Treatment with glucagon-like peptide-1 receptor agonists (GLP-1RAs), sodium glucose cotransporter- 2 (SGLT-2) inhibitors, and dipeptidyl peptidase 4 inhibitors (gliptins) unless stable for 120 days prior to screening or, if a historical biopsy is used, from 120 days prior to baseline liver biopsy until randomization.
* Use of concurrent medications prior to screening including:

  1. Anti-NASH therapy(s) including S-adenosyl methionine (SAMe), ursodeoxycholic acid (UDCA), and obeticholic acid in the period from 90 days prior to screening or, if a historical biopsy is used, from 90 days prior to baseline liver biopsy until randomization. For resmetirom; 120 days prior to screening or if a historical biopsy is used, from 120 days prior to baseline liver biopsy until randomization.
  2. Antidiabetic mediation which may impact NASH histology including thiazolidinediones (pioglitazone, rosiglitazone) in the period from 90 days prior to screening or, if a historical biopsy is used, from 90 days prior to baseline liver biopsy until randomization.
  3. Immune modulatory agents including anti-TNF-α therapies (infliximab, adalimumab, etanercept) or anti-integrin therapy (namixilab) in the period from 28 days prior to screening or if a historical biopsy is used from 28 days prior to baseline liver biopsy until randomization.
  4. Any treatment or anticipated initiation (intended use for more than 14 consecutive days) of medications known to have an effect on steatosis (e.g. treatment with corticosteroids [topical and inhaled are allowed]), methotrexate, tamoxifen, valproic acid, amiodarone or tetracycline, estrogens in doses higher than used in oral contraceptives, vitamin A, L-asparaginase, valproate, chloroquine, or antiretroviral drugs in the period from 28 days prior to screening or, if a historical biopsy is used, from 28 days prior to baseline liver biopsy until randomization.
  5. Treatment with orlistat, zonisamide, topiramate, phentermine, lorcaserin, bupropion, or naltrexone alone, or in combination or any other medication, that could promote weight loss, in the opinion of the investigator, in the period from 28 days prior to screening or if a historical biopsy is used from 28 days prior to baseline liver biopsy until randomization.
* Changing doses of statins (simvastatin, pitavastatin, pravastatin, atorvastatin, fluvastatin, lovastatin, rosuvastatin) or fibrates (clofibrate, Fenofibrate) in the 90 days preceding screening until randomization.
* Use of drugs that are known CYP2C8 inhibitors/substrate in the 28 days preceding screening until randomization.
* History of liver transplant
* Any weight reduction surgery in the 2 years prior to screening or planned during the study (weight reduction surgery is disallowed during the study), and malabsorptive weight loss surgery (Rouxen-Y or distal gastric bypass) at any time prior to screening.

Note: Lap banding, if the band has been removed >6 months before baseline liver biopsy, or intragastric balloon, if the balloon has been removed > 6 months before baseline liver biopsy, is allowed.

* Type 1 diabetes mellitus
* History of stomach or intestinal surgery or resection within the six months prior to screening that would potentially alter absorption and/or excretion of orally administered drugs as judged by the investigator.
* Unstable cardiovascular disease, including:

  1. unstable angina, (i.e., new or worsening symptoms of coronary heart disease) in the 90 days before screening and throughout the screening period; acute coronary syndrome in the 24 weeks before screening and throughout the screening period;
  2. acute myocardial infarction in the 90 days before screening and throughout the screening period; or heart failure of New York Heart Association class (III - IV), worsening congestive heart failure, or coronary artery intervention, in the 24 weeks before screening and throughout the screening period.
  3. history of unstable cardiac dysrhythmias
  4. uncontrolled hypertension at screening
  5. stroke or transient ischemic attack in the 24 weeks before screening
* History of myopathies or evidence of active muscle disease demonstrated by CPK ≥ 5 times ULN at screening.
* For subjects with elevated baseline ALT, AST, or ALP; ALT, AST, or ALP exceeding by more than 50% at Visit 2 reading compared to Visit 1 Note: If the ALT, AST or ALP values at Visit 2 exceed by more than 50% from Visit 1, then a third value will be measured to assess for the trend. If the third value shows continued increase ≥ 10%, then subject is considered ineligible for randomization.
* Any of the following laboratory values at screening:

  1. Hemoglobin <9 g/dL
  2. WBC count <2.5 × 103/µL
  3. Neutrophil count <1.5 × 103/µL
  4. Platelets <140 × 103/µL [if low platelet count is due to reasons other than liver disease as assessed by a hematologist, participants may be eligible if the platelet count is > 75 x 103/µL] as per investigator's discretion]
  5. INR ≥ 1.3 (in the absence of anticoagulants)
  6. Total bilirubin > ULN except in Gilbert's syndrome. In subjects with known Gilbert's syndrome, direct bilirubin > 2 x ULN
  7. Albumin <3.5 g/dL
  8. eGFR <60 mL/min/1.73 m2
  9. ALP ≥ 2x ULN
  10. ALT or AST ≥ 250 U/L
* Participation in any other therapeutic clinical study and on active treatment in the past 90 days of the screening.
* History of benign or malignant bladder tumors, and/or hematuria or has current hematuria except due to a urinary tract infection.
* History of malignancy in the past 5 years and/or active neoplasm with the exception of resolved superficial nonmelanoma skin cancer.
* Known allergy, sensitivity or intolerance to the study drug, comparator or formulation ingredients.
* Pregnancy-related exclusions, including:

  1. Pregnant/lactating female (including positive pregnancy test at screening)
  2. Pregnancy should be avoided by male and female participants either by true abstinence or the use of an acceptable effective contraceptive measures for the duration of the study and for at least 1 month after the end of the study treatment
* History or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for the study (such as poorly controlled psychiatric disease, HIV, coronary artery disease or active gastrointestinal conditions that might interfere with drug absorption)
* Receiving an elemental diet or parenteral nutrition.
* Chronic pancreatitis or pancreatic insufficiency.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Resolution of steatohepatitis with no worsening of fibrosis | 52 Weeks/EOT
  Resolution of steatohepatitis is defined as absent fatty liver disease or isolated or simple steatosis without steatohepatitis and a NAS of 0-1 for inflammation, 0 for ballooning, and any value for Steatosis

SECONDARY OUTCOMES:
Improvement in liver fibrosis with no increase in NAS for ballooning, inflammation or steatosis | Week 52/EOT
  Proportion of subjects achieving improvement in liver fibrosis (reduction of at least one stage) with no increase in NAS for ballooning, inflammation or steatosis
2 points improvement in NAS | Week 52/EOT
  Proportion of subjects with at least 2 points improvement in NAS at Week 52/EOT with at least 1-point improvement in either ballooning or inflammation and no worsening of liver fibrosis
Improvement in steatosis, ballooning, inflammation and fibrosis from liver biopsy | Week 52/EOT
  Proportion of subjects with ≥1 point improvement in steatosis, ballooning, inflammation and fibrosis
Decrease in SAF score on liver biopsy | Week 52/EOT
  Proportion of subjects with decrease in SAF score ≥2 combining hepatocellular inflammation and ballooning without worsening of fibrosis
Histological score changes in steatosis, ballooning, inflammation, and fibrosis | Week 52/EOT
  Change from baseline in steatosis, ballooning, inflammation, and fibrosis
Change in liver enzyme parameters including (ALT, AST, ALP, GGT, total bilirubin, albumin) | Week 52/EOT
  Change from baseline in liver enzyme parameters (ALT, AST, ALP, GGT, total bilirubin, albumin)
Change in non-invasive markers of steatosis | Week 52/EOT
  Change from baseline in non-invasive markers of steatosis (Enhanced Liver Fibrosis [ELF] test, Fibrosis 4 [FIB 4], APRI [AST to Platelet Ratio Index], NFS [NAFLD Fibrosis Score], PRO-C3)
Change in n lipid parameters including (TG, LDLC, TC, HDL-C, non-HDL-C, VLDL-C | Week 52/EOT
  Change from baseline in lipid parameters (TG, LDLC, TC, HDL-C, non-HDL-C, VLDL-C)
Change in body weight (any change from baseline) | Week 52/EOT
  Change from baseline in body weight
Change in insulin resistance marker, HOMA-IR | Week 52/EOT
  Change from baseline in insulin resistance marker (HOMA-IR)
Change in inflammatory markers including (CK-18 [M30], IL-6, CRP) | Week 52/EOT
  Change from baseline in inflammatory markers (CK-18 [M30], IL-6, CRP)
Change in glucose homeostasis markers including (HbA1c, FPG) | Week 52/EOT
  Change from baseline in glucose homeostasis markers (HbA1c, FPG)

CONTACTS AND LOCATIONS:
Overall Officials: Deven V. Parmar, MD, FCP, Study Director — Zydus Therapeutics Inc.
Locations (129):
- United States (101):
  - Zydus US032, Birmingham, Alabama
  - Zydus US079, Homewood, Alabama
  - Zydus US047, Phoenix, Arizona
  - Zydus US025, Tucson, Arizona
  - Zydus US087, Tucson, Arizona
  - Zydus US029, Tucson, Arizona
  - Zydus US118, Chula Vista, California
  - Zydus US041, Fresno, California
  - Zydus US111, Gardena, California
  - Zydus US013, Huntington Park, California
  - Zydus US065, La Jolla, California
  - Zydus US094, Lancaster, California
  - Zydus US080, Long Beach, California
  - Zydus US090, Long Beach, California
  - Zydus US022, Los Angeles, California
  - Zydus US062, Los Angeles, California
  - Zydus US023, Murrieta, California
  - Zydus US052, Orange, California
  - Zydus US012, Panorama City, California
  - Zydus US039, Aurora, Colorado
  - Zydus US122, Clearwater, Florida
  - Zydus US057, Fort Myers, Florida
  - Zydus US108, Hallandale, Florida
  - Zydus US096, Hialeah Gardens, Florida
  - Zydus US003, Lakeland, Florida
  - Zydus US016, Lakewood Rch, Florida
  - Zydus US125, Largo, Florida
  - Zydus US001, Maitland, Florida
  - Zydus US124, Maitland, Florida
  - Zydus US007, Miami, Florida
  - Zydus US024, Miami, Florida
  - Zydus US034, Miami, Florida
  - Zydus US038, Miami, Florida
  - Zydus US121, Miami, Florida
  - Zydus US054, Miami, Florida
  - Zydus US098, Miami Lakes, Florida
  - Zydus US099, Naples, Florida
  - Zydus US081, Ocala, Florida
  - Zydus US085, Orlando, Florida
  - Zydus US104, Port Orange, Florida
  - Zydus US004, Winter Park, Florida
  - Zydus US107, Dalton, Georgia
  - Zydus US113, Gainesville, Georgia
  - Zydus US114, Marietta, Georgia
  - Zydus US119, Savannah, Georgia
  - Zydus US020, Indianapolis, Indiana
  - Zydus US100, West Des Moines, Iowa
  - Zydus US049, Kansas City, Kansas
  - Zydus US071, Houma, Louisiana
  - Zydus US014, Marrero, Louisiana
  - Zydus US123, West Monroe, Louisiana
  - Zydus US017, Boston, Massachusetts
  - Zydus US092, Chesterfield, Michigan
  - Zydus US019, Wyoming, Michigan
  - Zydus US115, Saint Paul, Minnesota
  - Zydus US074, Columbia, Missouri
  - Zydus US120, Kansas City, Missouri
  - Zydus US116, Reno, Nevada
  - Zydus US077, Sparta, New Jersey
  - Zydus US069, Manhasset, New York
  - Zydus US066, New York, New York
  - Zydus US018, Asheville, North Carolina
  - Zydus US027, Charlotte, North Carolina
  - Zydus US010, Cincinnati, Ohio
  - Zydus US009, Cincinnati, Ohio
  - Zydus US035, Cleveland, Ohio
  - Zydus US072, Springboro, Ohio
  - Zydus US060, Hershey, Pennsylvania
  - Zydus US053, Philadelphia, Pennsylvania
  - Zydus US015, Charleston, South Carolina
  - Zydus US030, Charleston, South Carolina
  - Zydus US073, Columbia, South Carolina
  - Zydus US075, Greenwood, South Carolina
  - Zydus US112, Summerville, South Carolina
  - Zydus US011, Hermitage, Tennessee
  - Zydus US028, Nashville, Tennessee
  - Zydus US002, Arlington, Texas
  - Zydus US051, Austin, Texas
  - Zydus US101, Austin, Texas
  - Zydus US089, Bellaire, Texas
  - Zydus US105, Brownsville, Texas
  - Zydus US095, Edinburg, Texas
  - Zydus US106, Edinburg, Texas
  - Zydus US061, Fort Worth, Texas
  - Zydus US067, Houston, Texas
  - Zydus US109, Houston, Texas
  - Zydus US005, Houston, Texas
  - Zydus US110, Houston, Texas
  - Zydus US117, Katy, Texas
  - Zydus US031, San Antonio, Texas
  - Zydus US103, San Antonio, Texas
  - Zydus US036, San Antonio, Texas
  - Zydus US102, San Antonio, Texas
  - Zydus US043, San Antonio, Texas
  - Zydus US008, San Antonio, Texas
  - Zydus US078, Waco, Texas
  - Zydus US076, Wichita Falls, Texas
  - Zydus US088, Ogden, Utah
  - Zydus US070, Manassas, Virginia
  - Zydus US082, Richmond, Virginia
  - Zydus US021, Richmond, Virginia
- Argentina (13):
  - Zydus AR004, Buenos Aires
  - Zydus AR001, CABA
  - Zydus AR013, CABA
  - Zydus AR007, CABA
  - Zydus AR006, CABA
  - Zydus AR005, CABA
  - Zydus AR008, CABA
  - Zydus AR012, CABA
  - Zydus AR003, CABA
  - Zydus AR009, Mar del Plata
  - Zydus AR011, Mar del Plata
  - Zydus AR002, Ramos Mejía
  - Zydus AR010, Rosario
- Zydus US097, San Juan, Puerto Rico, Puerto Rico
- Turkey (Türkiye) (14):
  - Zydus TR003, Adana
  - Zydus TR002, Ankara
  - Zydus TR001, Ankara
  - Zydus TR004, Bursa
  - Zydus TR005, Gaziantep
  - Zydus TR009, Istanbul
  - Zydus TR008, Istanbul
  - Zydus TR007, Izmir
  - Zydus TR006, Izmir
  - Zydus TR011, Kayseri
  - Zydus TR010, Kocaeli
  - Zydus TR012, Mersin
  - Zydus TR013, Rize
  - Zydus TR014, Trabzon